CLINICAL TRIAL: NCT02148588
Title: How "Central" is Central Post-stroke Pain? Investigating the Role of Peripheral Sensory Input in Maintaining Central Pain
Brief Title: Peripheral Sensory Input in Central Post Stroke Pain (CPSP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Assistant Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201405121
Record Dates: First submitted 2014-05-15; First posted 2014-05-28 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Central Post Stroke Pain
Keywords: Central Post Stroke Pain; Nerve block
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pain testing (Experimental): Completion of NPSI questionnaire
  Sensory mapping of the affected limb
  Quantitative Sensory Testing
  Patients will have a peripheral nerve blockade
  Interventions: Drug: Ultrasound-guided peripheral nerve block with 2% lidocaine

INTERVENTIONS:
Drug: Ultrasound-guided peripheral nerve block with 2% lidocaine — Patients will have a peripheral nerve blockade with a local anesthetic (lidocaine)
  Assessment of spontaneous and evoked pain responses
  Completion of NPSI questionnaire
  Mapping of the affected limb

SUMMARY:
Prospective, open-label study in 10 patients with Central Post Stroke Pain (CPSP). The study will evaluate the effects of peripheral nerve blockade on spontaneous pain and evoked thermal and mechanical responses in CPSP, and assesses the associated local anesthetic pharmacokinetics.

ELIGIBILITY:
Each subject must meet all of the following criteria:

* Age ≥18;
* CPSP affecting an upper or a lower limb, in a distribution that may be completely covered by a peripheral nerve block;
* Patient fulfills all mandatory criteria for CPSP, fulfills at least one supportive criteria, and has definite CPSP by probability grading.
* Pain duration at least 3 months;
* Spontaneous pain intensity (average pain in past week) of ≥ 4 on 0-10 Numerical Rating Scale (NRS).

Exclusion Criteria

Subjects will not be enrolled if any of the following criteria exist:

* Not giving consent to participate in the study;
* Significant psychiatric or cognitive impairment;
* Moderate to severe renal or liver failure;
* Concomitant treatment with warfarin or other anticoagulants;
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12-15 (Actual); Study Completion 2017-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PHD, Principal Investigator — Washington Univesity School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- The Entire Cohort: All participants received a peripheral nerve block
Period: Overall Study
Arm/Group | The Entire Cohort
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | The Entire Cohort
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
  Denmark | 1

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Spontaneous Pain Intensity After a Peripheral Nerve Block.
Description: Reduction in spontaneous pain intensity in the painful extremity from baseline to 30 minutes after a peripheral nerve block.Spontaneous pain intensity was measured on 0-10 numerical rating scale (NRS), where 0 represents "no pain", and 10 represents "worst pain imaginable"
Time Frame: baseline and 30 minutes
Population: ITT
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | The Entire Cohort
Number analyzed (Participants) | 8
units on a scale
  Baseline pain intensity | 6.5 [4.3 to 7.0]
  Pain intensity after the block | 0.0 [0.0 to 0.0]

2. Secondary Outcome: Change in the Intensity of Cold Sensation
Description: The intensity of cold sensation (application of roller cooled down to 20 degrees Celsius) was measured on 0-10 scale, where 5 represents "normal" sensation (comparable to contralateral non-painful extremity). Higher scores indicate increased sensitivity (10= painful cold); lower scores represent reduced sensitivity (0=no cold sensation)
Time Frame: baseline and 30 min
Population: The entire cohort
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | The Entire Cohort
Number analyzed (Participants) | 8
units on a scale
  Baseline | 7 [4.5 to 7.8]
  30 min after the block | 0.0 [0.0 to 1.5]

3. Secondary Outcome: Change in the Intensity of Warm Sensation
Description: The intensity of warm sensation (application of roller heated up to 40 degrees Celsius) was measured on 0-10 scale, where 5 represents "normal" sensation (comparable to contralateral non-painful extremity). Higher scores indicate increased sensitivity (10= painful hot); lower scores represent reduced sensitivity (0=no warmth sensation)
Time Frame: baseline and 30 min
Population: The entire cohort
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Entire Cohort
Number analyzed (Participants) | 8
units on a scale
  Baseline | 5.9 (1.4)
  30 min after the block | 0.5 (1.1)

4. Secondary Outcome: Change in the Intensity of Pinprick Sensation
Description: The intensity of pinprick sensation (application of Semmes-Weinstein monofilament #6.1, ~100g target force) was measured on 0-10 scale, where 5 represents "normal" sensation (comparable to contralateral non-painful extremity). Higher scores indicate increased sensitivity (10= painful sharp); lower scores represent reduced sensitivity (0=no pricking sensation)
Time Frame: baseline and 30 min
Population: The entire cohort
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Entire Cohort
Number analyzed (Participants) | 8
units on a scale
  Baseline | 5.0 (2.1)
  30 min after block | 1.1 (2.2)

5. Secondary Outcome: Change in the Intensity of Brush Sensation
Description: The intensity of brush sensation (application of SENSELab Brush-05) was measured on 0-10 scale, where 5 represents "normal" sensation (comparable to contralateral non-painful extremity). Higher scores indicate increased sensitivity (10= painful brushing sensation); lower scores represent reduced sensitivity (0=no brushing sensation)
Time Frame: baseline and 30 min
Population: The entire cohort
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Entire Cohort
Number analyzed (Participants) | 8
units on a scale
  Baseline | 4.5 (1.9)
  30 min after block | 1.0 (1.4)

6. Secondary Outcome: Reported Pain/Dysesthesia Descriptors on NPSI Questionnaire
Description: Composite scores on NPSI (Neuropathic Pain Symptom Inventory) questionnaire before and 40 minutes after the peripheral nerve block.
  The NPSI assesses participant ranking of specific neuropathic pain descriptors, each ranked on a 0-10 scale, where 0 represents no burning/squeezing/electric shocks (etc), and 10 represents worst burning/squeezing/electric shocks (etc).
  The scores on individual questions are grouped (averaged) into the three following subscales (each subscale scores ranging from 0 to 10):
  * Burning pain
  * Paroxysmal pain
  * Paresthesia/dysesthesia
Time Frame: baseline and 40 min
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Entire Cohort
Number analyzed (Participants) | 8
units on a scale
  Burning pain- baseline | 4.1 (3.7)
  burning pain - 40 min after block | 0.0 (0.0)
  paroxysmal pain - baseline | 2.6 (2.1)
  Paroxysmal pain - 40 min after block | 0.0 (0.0)
  paresthesia/dysesthesia - baseline | 3.6 (3.3)
  paresthesia/dysesthesia - 40 min after block | 0.9 (1.3)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | The Entire Cohort
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Entire Cohort (N=8)
Perioral numbness (Nervous system disorders) | 2 (2) — Two patients reported perioral numbness for 14 and 10 minutes, respectively. Resolved spontaneously
Dizziness (Nervous system disorders) | 1 (1) — One subject reported dizziness (for 10 minutes), resolved spontaneously
Vasovagal response (Nervous system disorders) | 1 (1) — One patient experienced a vasovagal response during needle placement, but recovered uneventfully, and the study team proceeded with the block 5 minutes thereafter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No